CLINICAL TRIAL: NCT02855658
Title: Modulation of Immunity-related Gene Expression Under the Chinese Herbal Formula SS-1 Treatment for Sjögren's Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); China Medical University, China (Other); National Research Program for Biopharmaceuticals, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH105-REC3-025
Record Dates: First submitted 2016-07-13; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Sjögren's Syndrome
Keywords: Sjögren's syndrome; Gan-Lu-Yin; Sang-Ju-Yin; Xuefu-Zhuyu-Decoction; Oxidative stress; Immune regulation; Gene modulation; SS-1
MeSH Terms: conditions — Sjogren's Syndrome | interventions — sang ju yin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SS-1 (Experimental): SS-1 is composed of the powder of Gan-Lu-Yin, Sang-Ju-Yin and Xuefu-Zhuyu-Decoction with the ratio of 2:1:1. Patients take 6 gram of experiment medicine three times per day.
  Interventions: Drug: SS-1
- Placebo (Placebo Comparator): The placebo is composed of corn starch, pigment and minimal dose of 1% SS-1. Patients take 6 gram of experiment medicine three times per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SS-1 — The patients will be divided into two groups (A and B) at random and all of them keep the routine treatment in the rheumatology OPD. Group A patients will receive 12 weeks SS-1 treatment first, and then stop the SS-1 for 4 weeks for wash-out phase, and then receive 12 weeks placebo treatment. Group B patients receive 12 weeks placebo first, and then stop the placebo treatment for 4 weeks for wash-out phase, and then receive 12 weeks SS-1 treatment. SS-1 is composed of 3 traditional Chinese herbal formula: Gan-Lu-Yin, Sang-Ju-Yin and Xuefu-Zhuyu-Decoction with the ratio of 2:1:1. The placebo is composed with corn starch, pigment and minimal dose of 1% SS-1. Patients in both groups take 6 gram of SS-1/Placebo three times per day.
  Other Names: Gan-Lu-Yin, Sang-Ju-Yin and Xuefu-Zhuyu-Decoction
  Arms: SS-1
Drug: Placebo — The placebo is composed of corn starch, pigment and minimal dose of 1% SS-1. Patients take 6 gram of experiment medicine three times per day.
  Other Names: 1% SS-1
  Arms: Placebo

SUMMARY:
To evaluate the modulation of immunity-related gene expression for the Sjögren's syndrome under Chinese herbal medicine (SS-1) treatment.

DETAILED DESCRIPTION:
Objective: To evaluate the modulation of immunity-related gene expression for the Sjögren's syndrome under Chinese herbal medicine (SS-1) treatment.

Method:

The evidence of the regulation of oxidative-related cytokines and the antioxidant capacity could be provided from the previous randomized, double-blinded, placebo-controlled, cross-over design, two-center clinical trial for evaluating the effect of Chinese herbal medicine (SS-1) for the Sjögren's syndrome patients. However, the clinical trail could not find out the modulation of immunity-related gene expression for SS-1 treatment, and it did set up a healthy control group for SS-1 comparison. This study want to establish a healthy control group for evaluating the normal range of oxidative stress and cytokines, which this work could be used to compare with the 72 SS-1 subjects in previous study. And This study also want to analyze the 770 immunity-related gene expression for the Sjögren's syndrome under the SS-1 treatment: (1) The best 20 (at least) efficacy SJS subjects who were evaluated before and after SS-1 treatments. (2) The 10 (at least) healthy control subjects. The findings could provide the evidence on the modulation of immunity-related gene expression for clinical manifestation, oxidative stress and cytokine in Sjögren's syndrome patients.

Expected Results:

1. Establish the normal range of oxidative stress and cytokines for healthy control group.
2. To evaluate the regulatory effect on oxidative stress and cytokine secretion between SS-1 group and healthy control group.
3. To evaluate the immunity-related gene expression for the Sjögren's syndrome under the SS-1 treatment.
4. To evaluate the immunity-related gene expression among the best efficacy SJS subjects and healthy control subjects.
5. To evaluate the immunity-related gene expression with the characteristic of TCM tongue diagnosis.
6. To analyze the correlation among clinical manifestations, Sjögren's syndrome -related clinical questionnaires and immunity-related gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Primary or Secondary Sjögren's syndrome patient
* Age from 20 to 75 year old, male or female patient
* Fit the criteria of 2002 year American-European classification
* If the subject took Cyclosporine, Cevimeline, Pilocarpine, Rituximab or other biological agent before enter into our study, the subject need to stop these drugs for one month
* If the subject took Gan-Lu-Yin, Sang- Ju-Yin or Xuefu-Zhuyu-Decoction before enter into our study, the subject need to stop these drugs for one month
* Secondary Sjögren's syndrome patient:

  * Stable treatment: Steroid (≦10mg/d) and fixed hydroxychloroquine dose before 3 months enrolled
  * No abnormal change of immunology, liver, kidney, and blood function
  * No major life threatened condition

Exclusion Criteria:

* Alcohol abuse, DM (Glucose PC>200mg/dL) and major life threatened condition
* Pregnancy or breast feeding
* Abnormal liver and kidney function
* Forbid steroid pulse therapy before 3 months enrolled into our study, and forbid the Chinese herbal medicine except SS-1

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Ocular surface disease index (OSDI) | 7 months
  OSDI is an questionnaire of dry eye.
EULAR Sjogren's syndrome patient reported index (ESSPRI) | 7 months
  ESSPRI is an questionnaire of dry, pain and fatigue.
Sjogren's syndrome symptoms Questionnaire | 7 months
  Sjogren's syndrome symptoms Questionnaire is an questionnaire of dry month.
Schirmer's test | 7 months
  Schirmer's test is an objective detection of dry eye, which this test use paper strips inserted into the eye for 5 minutes to measure the production of tears.
Salivary scintigraphy | 7 months
  Salivary scintigraphy is an objective detection of dry month, which is used to detect the salivary flow in parotid gland of Sjogren's syndrome.

SECONDARY OUTCOMES:
Oxidative stress and antioxidant capacity | 7 months
  To evaluate the effect of the SS-1 on the oxidative stress and antioxidant capacity. The "relative ratio" is the unit of these biomarkers for oxidative stress and antioxidant capacity
Quality of life (SF-36) | 7 months
Regulatory effect on cytokine | 7 months
  To evaluate the effect of the SS-1 on the cytokine. The "pg/ml" is the unit of these biomarkers for oxidative stress and antioxidant capacity
Nanostring nCounter immune Panel | 7 months
  To evaluate the effect of the SS-1 on the immunity-related gene expression. Nanostring nCounter immune Panel is a tool for detecting the immunity-related gene expression.

OTHER OUTCOMES:
Adverse effect (AE) and Adverse drug reaction(ADR) | 7 months
  Monitor the Adverse effect (AE) and Adverse drug reaction(ADR) during the SS-1 trial.
Liver, Kidney and Blood function monitor | 7 months
  Monitor the Liver, Kidney and Blood function monitor (RBC, WBC, Hb, Platelet, AST, ALT, BUN, Cre) of patient during the SS-1 trial, and the different units are listed below: WBC (1000/uL), RBC (million/uL), Hb (g/dL), Platelet (1000/uL), AST (U/L), ALT (U/L), BUN (mg/dL), Serum Creatinine (mg/dL).
Traditional Chinese medicine (TCM) tongue diagnosis | 7 months
  To evaluate the effect of the SS-1 on the TCM tongue diagnosis before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hen-Hong Chang, M.D., Ph.D., Study Chair — China Medical University Hospital
Locations (2):
- Taiwan (2):
  - Taoyuan Chang Gung Memorial Hospital, Gueishan Township, Taiwan
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chang CM, Chu HT, Wei YH, Chen FP, Wang S, Wu PC, Yen HR, Chen TJ, Chang HH. The Core Pattern Analysis on Chinese Herbal Medicine for Sjogren's syndrome: A Nationwide Population-Based Study. Sci Rep. 2015 Apr 29;5:9541. doi: 10.1038/srep09541. Erratum In: Sci Rep. 2015 Oct 08;5:14887. doi: 10.1038/srep14887. Sci Rep. 2017 May 25;7:46824. doi: 10.1038/srep46824. PMID 25923413
- See also: NCT02110446: Evaluation of the Efficacy and the Mechanism of Chinese Herbal Formula SS-1 for Sjögren's Syndrome (SS-1) — https://clinicaltrials.gov/ct2/show/study/NCT02110446